CLINICAL TRIAL: NCT06502145
Title: Iadademstat With Hypomethylating Agent in Patients With Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Guru Subramanian Guru Murthy, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00053184
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose level -1 (Experimental): Dose level -1 will be considered only if there are dose-limiting toxicities at dose level 0. This is a regimen of azacitidine and iadademstat.
  Interventions: Drug: Azacitidine Level -1; Drug: Iadademstat Level -1
- Dose level 0 (Experimental): This is a regimen of azacitidine and iadademstat.
  Interventions: Drug: Azacitidine Level 0; Drug: Iadademstat Level 0
- Dose level 1 (Experimental): This is a regimen of azacitidine and iadademstat.
  Interventions: Drug: Azacitidine Level 1; Drug: Iadademstat Level 1
- Maximum Tolerated Dose (MTD) (Experimental): The MTD is the highest dose level at which no more than 1 of 6 treated participants, experiences a dose-limiting toxicity.
  Interventions: Drug: Iadademstat Level -1; Drug: Iadademstat Level 0; Drug: Iadademstat Level 1

INTERVENTIONS:
Drug: Azacitidine Level -1 — Intravenous (IV) or subcutaneous (SC) 75 mg / m^2 days 1-7 X 28 days.
  Other Names: Vidaza; Onureg
  Arms: Dose level -1
Drug: Azacitidine Level 0 — Intravenous (IV) or subcutaneous (SC) 75 mg / m^2 days 1-7 X 28 days.
  Other Names: Vidaza; Onureg
  Arms: Dose level 0
Drug: Azacitidine Level 1 — Intravenous (IV) or subcutaneous (SC) 75 mg / m^2 days 1-7 X 28 days.
  Other Names: Vidaza; Onureg
  Arms: Dose level 1
Drug: Iadademstat Level -1 — 75 µg by mouth (PO) 5 days on, 2 days off for 2 weeks every 28 days.
  Arms: Dose level -1; Maximum Tolerated Dose (MTD)
Drug: Iadademstat Level 0 — 75 µg PO 5 days on, 2 days off for 3 weeks every 28 days.
  Arms: Dose level 0; Maximum Tolerated Dose (MTD)
Drug: Iadademstat Level 1 — 100 µg PO 5 days on, 2 days off for 3 weeks every 28 days.
  Arms: Dose level 1; Maximum Tolerated Dose (MTD)

SUMMARY:
This is a phase I study with a primary objective of determining the recommended phase II dose of iadademstat with azacitidine in adult subjects with myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
This is a single-arm, open-label phase 1 study designed to evaluate the safety of iadademstat with azacitidine therapy. The trial will follow a 3+3 phase 1 dose-escalation design.

First, three participants are given a low dose of the experimental treatment and monitored for pre-specified toxicity events. If 0 participants experience one of these toxicity events, then the next group of three participants is enrolled at a higher dose. If two or three participants experience toxicity, then the next group of three participants is enrolled at a lower dose (or the study ends). If one participant experiences toxicity, another group of three participants is enrolled at the same dose (hence the name, 3+3): if one or more of those participants experience toxicity, then the dose is lowered for the next group of the study ends. Otherwise, if 0 of the additional participants experience toxicity, the next group is enrolled at a higher dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years or older.
2. Patients must have a diagnosis of myelodysplastic syndrome (MDS), or MDS / myeloproliferative neoplasm (MPN), chronic myelomonocytic leukemia (CMML) as defined by the World Health Organization (WHO) criteria.
3. Intermediate, high, or very-high risk by the Revised International Prognostic Scoring System (IPSS-R).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (0-3 if performance status is considered due to MDS).
5. Patient must have a body weight of at least 50 kg.
6. Patient must meet the following screening clinical laboratory values as specified below:

   a. Hematologic: white blood cell (count) (WBC) below 30 x 109/L. Hydroxyurea can be used to achieve this level b. Hepatic: i. Total bilirubin ≤1.5 x upper limit of normal (ULN). Patients with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits.

   ii. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x ULN.

   c. Renal: Serum creatinine ≤1.5 x ULN.
7. Patient is able to swallow oral medications.
8. Female subjects who:

   1. Are postmenopausal for at least one year before the screening visit, OR
   2. Are surgically sterile, OR
   3. If they are of childbearing potential:

   i. Agree to practice one highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through six months after the last dose of study drug (female and male condoms should not be used together), OR ii. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception).

   iii. Agree to not to donate or freeze egg(s) during the course of this study or within 180 days after receiving their last dose of study drug.
9. Male subjects, even if surgically sterilized (i.e., status post vasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study treatment period from the time of signing the informed consent through and through six months after the last dose of study drug (female and male condoms should not be used together), OR
   2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
   3. Agree to not to donate or freeze sperm during the course of this study or within 180 days after receiving their last dose of study drug.
10. Ability to provide informed consent or have a legally authorized representative provide consent.

Exclusion Criteria:

A potential study subject who meets any of the following exclusion criteria is ineligible to participate in the study:

1. Prior therapy with hypomethylating agent or Lysine-specific histone demethylase 1A (LSD1) inhibitor. If patients were treated with any other agents having KDM1A/LSD1 inhibitory activity (such as tranylcypromine or phenelzine or similar drugs), they are only allowed if treatment finalized at least 3 weeks prior to first dose on study.
2. Patient will require treatment while on study with concomitant drugs that target the 5- hydroxytryptamine2B (5-HT2B) receptor or the sigma nonspecific receptor (e.g., escitalopram, fluoxetine, sertraline) except for drugs that are considered absolutely essential for the care of the patient and with appropriate treatment monitoring.
3. Treatment with systemic antineoplastic chemotherapy within 14 days or 5 half-lives from the last dose - whichever is sooner - before Cycle 1, Day 1 of therapy. Radiation within 14 days before Cycle 1, Day 1 of therapy. The use of hydroxyurea for leukoreduction is permitted. Similarly, prior ESA, luspatarcept, or lenalidomide is allowed. Subjects must have recovered from the side effects of prior therapy per the treating physician's discretion.
4. Patient is on treatment with any investigational products within 3 weeks prior to the first dose of study treatment.
5. Patient has had major surgery within 4 weeks prior to the first study dose.
6. Patients with uncontrolled hypertension (i.e., systolic blood pressure >180 mm Hg, diastolic blood pressure >95 mm Hg). Use of anti-hypertensive agents to control hypertension before Cycle 1, Day 1 is allowed.
7. Patients with known poorly controlled diabetes (glycosylated hemoglobin (HbA1c) ≥8%) unless actively managed with appropriate therapy; patients with a history of transient glucose intolerance due to corticosteroid administration may be enrolled in this study if all other inclusion/exclusion criteria are met.
8. Patient has known active congestive heart failure New York Heart Association (NYHA) class 3 or 4 or patients with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 1 month prior to study entry demonstrates a left ventricular ejection fraction that is ≥40%.
9. Patients with known long QT Syndrome at screening.
10. History of allogeneic stem cell transplantation or CAR-T therapy within past 60 days.
11. Patient has evidence of active uncontrolled viral, bacterial, or systemic fungal infection (i.e., no signs of severe systemic inflammatory response that makes patient clinically unstable in the opinion of the investigator, and patient is hemodynamically stable, with sustained body temperature under 38°C for 48-72 hours before starting study treatment and does not need oxygen supplementation or pressors to maintain blood pressure). Patients with uncontrolled infection shall not be enrolled until the infection is treated and brought under control.
12. Manifestations of malabsorption due to prior gastrointestinal (GI) surgery or GI disease that may alter the absorption of iadademstat.
13. Pregnant or lactating / breastfeeding women.
14. Patient has any condition which, in the investigator's opinion, makes the patient unsuitable for study participation. For example, any inter-current illness or social situation that will limit compliance with study requirements. Any serious underlying medical or psychiatric condition (e.g., alcohol or drug abuse), dementia or altered mental status or any issue that would impair the ability of the patient to understand the informed consent form or that in the opinion of the investigator would contraindicate the patient's participation in the study or confound the results of the study.
15. Patient presents a known contraindication to any of the treatment drug excipients.
16. Patient has known active hepatic disorder or is known to be positive for hepatitis B or C infection with the exception of those with undetectable viral load within 3 months (Hepatitis B or C testing is not required for eligibility assessment).
17. Patient is known to have human immunodeficiency virus infection. (HIV testing is not required for eligibility assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of Iadademstat. | Up to two years
  The dose identified in this trial that will be used in future clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Guru Subramanian Guru Murthy, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No